CLINICAL TRIAL: NCT05176405
Title: Using Entertainment Media to Deliver Educational Messages About Mammography in Saudi Arabia
Brief Title: Entertainment Media to Deliver Educational Messages About Mammography in Saudi Arabia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: MCC-21-18633; HM20022255 (Other: Virginia Commonwealth University)
Record Dates: First submitted 2021-10-29; First posted 2022-01-04 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-08

CONDITIONS: Breast Cancer; Behavior
Keywords: Mammogram; Prevention
MeSH Terms: conditions — Breast Neoplasms; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Elissa's EE Song (Experimental): Participants will have to click on the watch button to start the YouTube video as it is without manipulation. Right after exposure, the first and second arms will be asked if they have seen either of the presented materials before.
  Interventions: Behavioral: You-Tube Video: Elissa's EE song
- Standard of Care (Active Comparator): Participants will be assigned to read general infographic messages adopted from the Saudi Ministry of Health (MOH) in the breast cancer early screening context in Arabic/English. Right after exposure, the first and second arms will be asked if they have seen either of the presented materials before.
  Interventions: Behavioral: Active Comparator: Standard of Care
- Control Group (No Intervention): The third arm of this trial is the control group who will not be exposed to any preventative messages.

INTERVENTIONS:
Behavioral: You-Tube Video: Elissa's EE song — Watch You-Tube video utilizing Entertainment-Education communication strategy.
  Arms: Elissa's EE Song
Behavioral: Active Comparator: Standard of Care — Reading materials containing information about early breast cancer screening in the form of infographics. Information is adopted from the Saudi Ministry of Health (MOH).
  Arms: Standard of Care

SUMMARY:
This clinical trial aims to test if Elissa's Entertainment-Education (EE) song can influence Saudi females' intention to perform breast cancer early screening via mammogram.

DETAILED DESCRIPTION:
This study will be guided by a scarcely applied theoretical model that integrates the issue involvement concept into the Theory of Planned Behavior (TPB) to test the role of issue involvement in predicting intention to perform breast cancer early screening via mammogram among Saudi females after exposure to EE message.

ELIGIBILITY:
Inclusion Criteria:

* Saudi Arabian
* female

Exclusion Criteria:

* Females 39 or younger
* females above age 69 years
* females who have had breast cancer
* females that have had risk-reducing bilateral mastectomies

Ages: 40 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-03-14 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
Measure the role of issue involvement in predicting intention to perform breast cancer early screening via mammogram among Saudi females after exposure to EE message. | 1 Day
  Right after exposure to the intervention, the first and second arms will be asked if they have seen either of the presented materials before. During the statistical analysis, the researcher will control for those who indicate seeing either of these materials. The three arms will be given one validated questionnaire that measures issue involvement (INV) and Theory of Planned Behaviors (TPB's) constructs. Issue involvement will be measured using a personal involvement inventory scale. Issue involvement will be answered on a 7-point Likert scale ranging from 1 (Not at all) to 7 (Very much) with six items: important, relevant, interesting, means a lot to me, valuable, and involving. The minimum value is 6 and the maximum value is 42. High scores mean a high level of involvement with mammography.

SECONDARY OUTCOMES:
Measure the Theory of Planned Behavior (TPB) construct attitude, to predict Saudi females' intention to perform breast cancer early screening via mammogram | 1 Day
  Attitude toward mammography will be measured directly by asking participants to indicate their level of agreement with the following three statements 1) Getting a mammogram in the next two years would be good; 2) Getting a mammogram in the next two years would be useful; and 3) Getting a mammogram in the next two years would be safe. The scores will be added together to measure Saudi females' attitudes toward mammography The minimum value is 3, and the maximum value is 15. A high score indicates a more positive attitude towards mammography.
Measure the TPB construct, subject norm, to predict Saudi females' intention to perform breast cancer early screening via mammogram | 1 day
  Subject norms will be measured utilizing the Theory of Planned Behavior Questionnaire. Subjective norms will be measured directly by asking participants to indicate their level of agreement with the following three statements 1) Most people who are important to me think I should get a mammogram in the next two years; 2) Most people who are important to me expect me to get a mammogram in the next two years; and 3) Most people who are important to me would approve of me getting a mammogram in the next two years The minimum value is 3 and the maximum value is 15. A high score indicates a more positive attitude towards mammography.
Measure the TPB construct perceived behavioral control, to predict Saudi females' intention to perform breast cancer early screening via mammogram | 1 day
  Perceived behavioral control will be measured directly by asking participants to indicate their level of agreement with the following three statements: 1) Whether or not I get a mammogram in the next two years is entirely up to me; 2) I believe it is feasible to get a mammogram in the next two years; and 3) I am confident that if I wanted I would be able to get a mammogram in the next two years. The scores will be added together to measure how much control do Saudi females have to perform mammography in the next two years. The expected minimum value is 3, while the maximum value is 15. A high score implies higher behavioral control toward mammography.
Compare the differences between EE viewers and non EE viewers in terms of issue involvement | 1 Day
  Involvement is measured utilizing the results from the personal involvement inventory scale (PII) scale. Issue involvement will be answered on a 7-point Likert scale ranging from 1 (Not at all) to 7 (Very much) with six items: important, relevant, interesting, means a lot to me, valuable, and involving. The expected minimum value is 6, while the maximum value of 42 with high scores implies a high level of involvement with the mammography.
Compare the differences between EE viewers and none EE viewers in terms of attitude. | 1 Day
  Attitude is measured directly by asking participants to indicate their level of agreement with the following three statements 1) Getting a mammogram in the next two years would be good; 2) Getting a mammogram in the next two years would be useful; and 3) Getting a mammogram in the next two years would be safe. The scores will be added together to measure Saudi females' attitudes toward mammography. The expected minimum value is 3, while the maximum value is 15. A high score means a more positive attitude toward mammography
Compare the differences between EE viewers and none EE viewers in terms of perceived behavioral control. | 1 Day
  Perceived behavioral control will be measured directly by asking participants to indicate their level of agreement with the following three statements: 1) Whether or not I get a mammogram in the next two years is entirely up to me; 2) I believe it is feasible to get a mammogram in the next two years; and 3) I am confident that if I wanted I would be able to get a mammogram in the next two years. The scores will be added together to measure how much control do Saudi females have to perform mammography in the next two years. The expected minimum value is 3, while the maximum value is 15. A high score implies higher behavioral control toward mammography.
Measure intention toward mammography | 1 Day
  Intention toward mammography will be measured directly by asking participants to indicate their level of agreement with the following three statements 1) I plan to get a mammogram in the next two years; 2) I want to get a mammogram in the next two years; 3) I will try to get a mammogram in the next two years. The scores will be added together to measure Saudi females' intention to perform mammography in the next two years. The expected minimum value is 3, while the maximum value is 15. A high score reflects stronger intentions toward mammography

CONTACTS AND LOCATIONS:
Overall Officials: Jeanine Guidry, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Currently there are no plans to make individual participant data (IPD) available to other researchers.